CLINICAL TRIAL: NCT05460416
Title: A Prospective Interventional Randomized Controlled Trial to Assess the Effect of Low Dose Acetylsalicylic Acid As a Preventive Treatment of Pre-eclampsia in Pregnant Women Who Underwent Frozen Embryo Transfer
Brief Title: Treatment Preventive for Pre-eclampsia by Acetylsalicylic Acid in Women Who Underwent Frozen Embryo Transfer
Acronym: TePPAFET
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Responsible Party: Principal Investigator, Julie Collee, Doctor, specialist in Obstetrics and Reproductive Medicine, Centre Hospitalier Régional de la Citadelle
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021/392; 2024-516816-72-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-11; First posted 2022-07-15 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Embryo Transfer; Hypertension, Pregnancy Induced
Keywords: embryo transfer; Hypertension, Pregnancy induced
MeSH Terms: conditions — Hypertension, Pregnancy-Induced | interventions — Aspirin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment by acetylsalicylic acid (Experimental)
  Interventions: Drug: Acetylsalicylic acid
- No treatment (No Intervention)

INTERVENTIONS:
Drug: Acetylsalicylic acid — 160mg once a day
  Arms: Treatment by acetylsalicylic acid

SUMMARY:
Title: A prospective multicentric interventional randomized controlled trial to assess the effect of low dose acetylsalicylic acid as a preventive treatment of pre-eclampsia in pregnant women who underwent frozen embryo transfer

DETAILED DESCRIPTION:
Method: Prospective, interventional, multicentric randomized controlled trial, to evaluate the utility of a preventive treatment with low dose acetylsalicylic acid from the embryo transfer and throughout pregnancy in patients who have had a frozen embryo transfer.

During the first consultation, patients will be introduced to the study. They can choose to participate or not. If they agree to participate, they will be randomized in two groups (1:1), treated or not. The randomization will be realized by the RedCap software. Patients with natural and modified natural cycle and hormone replacement treatment (HRT) cycle will be included. As soon as an evolutive intrauterine pregnancy is diagnosed, in the treated group, she will receive a daily dose of 160mg acetylsalicylic acid, until 36 weeks of amenorrhea. Patients of both groups will be followed twice a month (regular prenatal visit and phone call).

Primary goal: To assess the incidence of pre-eclamspia in women who underwent a frozen embryo transfer treated with 160mg of acetylsalicylic acid versus no treatment.

Primary endpoint: Mean number of women suffering from preeclampsia in the treated and not treated groups.

Secondary goals:

* To assess the incidence of pre-eclampsia in women who underwent a frozen embryo transfer in natural and modified natural cycle treated with 160mg acetylsalicylic acid versus without treatment Secondary Endpoint 1: mean number of women suffering from pre-eclampsia in treated and without treatment groups in women in natural and modified natural cycle
* To assess the incidence of pre-eclampsia in women who underwent a frozen embryo transfer in HRT cycle treated with 160mg acetylsalicylic acid versus without treatment Secondary Endpoint 2: mean number of women suffering from pre-eclampsia in treated and without treatment groups in women in HRT cycle
* To assess the number of miscarriage in frozen embryo transfer with natural and modified natural cycle and with HRT cycle.

Secondary Endpoint 3: mean number of miscarriage

- To assess the number of pre-eclampsia in frozen embryo transfer with natural and modified natural cycle and with HRT cycle.

Secondary Endpoint 4: mean number of pre-eclampsia

Duration: the study duration for the participant will be maximum 12 months (from inclusion before embryo transfer until delivery). The total duration study will be maximum 4 years from the first patient first inclusion visit until the last visit of study patient.

Number of participants: 120 patients per group, HRT cycle versus without treatment, spontaneous cycle vs without treatment. Due to miscarriage risk, a total of 276 women will be enrolled.

Inclusion criteria:

* Healthy women from [18 - 43] years-old, planned for a frozen embryo transfer, with natural and modified natural or HRT cycle
* Who have given their informed consent
* Who have a confirmed pregnancy at week 6 of amenorrhea.

Exclusion criteria

* Women presenting one risk factor for preeclampsia: multiple pregnancy, history of preeclampsia, BMI > 30, lupus syndrome, preexistent proteinuria, non-treated chronic high blood pressure (>140/90), antiphospholipid antibody syndrome, diabetes (fasting blood sugar >126mg/dl)
* Contraindication to acetylsalicylic acid (at risk of active hemorrhage (like hemophilia, …); at risk of or who have a gastro-duodenal ulcer; at risk or how have a terminal renal or hepatic in-sufficiency (only if acetylsalicylic acid is given at high dose)
* Already treated with acetylsalicylic acid
* Treatment with anticoagulants or non-steroid anti-inflammatory drugs

ELIGIBILITY:
Inclusion Criteria:

* Healthy women from [18 - 43] years-old, planned for a frozen embryo transfer, with natural and modified natural or HRT cycle
* Who have given their informed consent
* Who have a confirmed pregnancy at week 6 of amenorrhea.

Exclusion Criteria:

* Women presenting one risk factor for preeclampsia: multiple pregnancy, history of preeclampsia, BMI > 30, lupus syndrome, preexistent proteinuria, non-treated chronic high blood pressure (>140/90), antiphospholipid antibody syndrome, diabetes (fasting blood sugar >126mg/dl)
* Contraindication to acetylsalicylic acid (at risk of active hemorrhage (like hemophilia, …); at risk of or who have a gastro-duodenal ulcer; at risk or how have a terminal renal or hepatic in-sufficiency (only if acetylsalicylic acid is given at high dose)
* Already treated with acetylsalicylic acid
* Treatment with anticoagulants or non-steroid anti-inflammatory drugs

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 276 (Estimated)
Dates: Start 2022-10-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean number of women suffering from pre-eclampsia in the treated and not treated groups. | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Henry, Principal Investigator — Centre Hospitalier Régional de la Citadelle
Locations (1):
- Centre Hospitalier Universitaire de Liège site Citadelle, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No